CLINICAL TRIAL: NCT05020249
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study to Evaluate the Efficacy and Safety of Bimekizumab in Adult Korean Study Participants With Moderate to Severe Plaque Psoriasis
Brief Title: A Study to Evaluate the Efficacy and Safety of Bimekizumab in Adult Korean Study Participants With Moderate to Severe Plaque Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PS0032
Record Dates: First submitted 2021-08-20; First posted 2021-08-25 (Actual); Results first posted 2024-03-22 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Moderate to Severe Plaque Psoriasis
Keywords: Moderate to Severe Plaque Psoriasis; Korean Study Participants; BKZ; UCB4940
MeSH Terms: interventions — bimekizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bimekizumab arm (Experimental): Study participants randomized to this arm will receive bimekizumab (BKZ; UCB4940) at pre-specified time points during the Treatment Period.
  Interventions: Drug: bimekizumab
- Placebo arm (Placebo Comparator): Study participants randomized to this arm will receive placebo (PBO) at pre-specified time points during the Treatment Period.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: bimekizumab — Study participants will receive bimekizumab administered through subcutaneous injection in a pre-specified sequence during the Treatment Period.
  Other Names: BKZ; UCB4940
  Arms: Bimekizumab arm
Other: Placebo — Study participants will receive placebo administered through subcutaneous injection in a pre-specified sequence during the Treatment Period.
  Other Names: PBO
  Arms: Placebo arm

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of bimekizumab compared with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Study participant must be at least 19 years of age at the time of signing the informed consent
* Study participant must be a Korean adult with a diagnosis of moderate to severe psoriasis (PSO)
* Study participant must have had plaque PSO for at least 6 months prior to the Screening Visit
* Study participant must have Psoriasis Area and Severity Index (PASI) ≥12 and body surface area (BSA) affected by PSO ≥10% and Investigator's Global Assessment (IGA) score ≥3 on a 5-point scale
* Study participant must be a candidate for systemic PSO therapy and/or phototherapy
* Study participant agrees not to change their usual sun exposure during the course of the study and to use ultraviolet A/ultraviolet B sunscreens if unavoidable exposure occurs
* A female study participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:
* Not a female of childbearing potential (FOCBP) OR A FOCBP who agrees to follow the contraceptive guidance during the Treatment Period and for at least 20 weeks after the last dose of study treatment

Exclusion Criteria:

* Subject has an active infection (except common cold), a serious infection, or a history of opportunistic or recurrent chronic infections
* Subject has concurrent acute or chronic viral hepatitis B or C or human immunodeficiency virus (HIV) infection
* Subject has known tuberculosis (TB) infection, is at high risk of acquiring TB infection, or has current or history of nontuberculous mycobacterium (NTMB) infection
* Subject has any active malignancy or history of malignancy within 5 years prior to the Screening Visit EXCEPT treated and considered cured cutaneous squamous or basal cell carcinoma, or in situ cervical cancer
* Study participant has a presence of active suicidal ideation or positive suicide behavior
* Study participant has a presence of moderately severe major depression or severe major depression
* Subject has a known hypersensitivity to any excipients of bimekizumab
* Subject has any other condition, including medical or psychiatric, which, in the Investigator's judgment, would make the subject unsuitable for inclusion in the study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2021-09-27 (Actual); Primary Completion 2022-09-05 (Actual); Study Completion 2022-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273
Locations (9):
- South Korea (9):
  - Ps0032 20211, Bucheon-si
  - Ps0032 20214, Busan
  - Ps0032 20215, Gwangju
  - Ps0032 20208, Seongnam-si
  - Ps0032 20210, Seongnam-si
  - Ps0032 20104, Seoul
  - Ps0032 20138, Seoul
  - Ps0032 20213, Seoul
  - Ps0032 20216, Seoul

IPD SHARING:
Plan to Share IPD: Yes
Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized individual patient-level data and redacted trial documents which may include: analysis-ready datasets, study protocol, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a prespecified time, typically 12 months, on a password protected portal. This plan may change if the risk of re-identifying trial participants is determined to be too high after the trial is completed; in this case and to protect participants, individual patient-level data would not be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: http://www.Vivli.org

REFERENCES:
- [Result] Youn SW, Jo SJ, Park CJ, Kim DH, Shin BS, Jeong KH, Bang CH, Cross N, Thirlwell J, Hoepken B. Bimekizumab efficacy and safety in Korean patients with moderate to severe plaque psoriasis: A phase 3, randomized, placebo-controlled, double-blinded study. J Dermatol. 2024 Nov;51(11):1392-1403. doi: 10.1111/1346-8138.17446. Epub 2024 Sep 27. PMID 39328126

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll study participants in September 2021 and concluded in September 2022.
Pre-assignment Details: The Participant Flow refers to the Randomized Set.
Groups:
- Placebo: Participants received placebo matched to bimekizumab subcutaneous (sc) injection every 4 weeks (Q4W) until Week 16. Placebo was used to maintain the blinding and is a real comparator in this study.
- Bimekizumab 320 mg Q4W: Participants received bimekizumab 320 milligrams (mg) sc injection Q4W until Week 16.
Period: Overall Study
Arm/Group | Placebo | Bimekizumab 320 mg Q4W
Started | 15 | 32
Completed | 14 | 32
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Randomized Set which consisted of all randomized study participants.
Groups:
- Placebo: Participants received placebo matched to bimekizumab sc injection Q4W until Week 16. Placebo was used to maintain the blinding and is a real comparator in this study.
- Bimekizumab 320 mg Q4W: Participants received bimekizumab 320 mg sc injection Q4W until Week 16.
- Total: Total of all reporting groups
Arm/Group | Placebo | Bimekizumab 320 mg Q4W | Total
Number analyzed (Participants) | 15 | 32 | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 32 | 47
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.2 (11.3) | 39.7 (9.0) | 39.9 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 9
  Male | 12 | 26 | 38
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 15 | 32 | 47
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 15 | 32 | 47

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Psoriasis Area and Severity Index 90 (PASI90) Response at Week 16
Description: The PASI90 response assessments are based on a 90% improvement in the PASI score from Baseline. This is a scoring system that averages the redness, thickness, and scaliness of the psoriatic lesions (on a 0-4 scale), and weights the resulting score by the area of skin involved. Body divided into 4 areas: head, arms, trunk to groin, and legs to top of buttocks. Assignment of an average score for the redness, thickness, and scaling for each of the 4 body areas with a score of 0 (clear) to 4 (very marked). Determining the percentage of skin covered with PSO for each of the body areas and converting to a 0 to 6 scale. Final PASI= average redness, thickness, and scaliness of the psoriatic skin lesions, multiplied by the involved psoriasis area score of the respective section, and weighted by the percentage of the person's affected skin for the respective section. The minimum possible PASI score is 0= no disease, the maximum score is 72= maximal disease.
Time Frame: Week 16
Population: Randomized Set consisted of all randomized study participants. Study participants with an intercurrent event (discontinuation of IMP prior to Week 16) or who had missing data at Week 16 are counted as non-responders (Non responder imputation (NRI)).
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Bimekizumab 320 mg Q4W
Number analyzed (Participants) | 15 | 32
percentage of participants | 0 | 81.3
Statistical Analysis 1: Comparison: Placebo vs Bimekizumab 320 mg Q4W; Test type: Superiority; p < 0.001, Fisher Exact — P-values for the comparison of treatment groups are based on the Fisher's exact test

2. Primary Outcome: Percentage of Participants With an Investigator's Global Assessment (IGA) 0/1 (Clear or Almost Clear With at Least 2-category Improvement From Baseline) Response at Week 16
Description: The Investigator's Global Assessment measures the overall psoriasis severity following a 5-point scale (0-4), where scale 0= Clear, no signs of psoriasis; post-inflammatory hyperpigmentation may be present, scale 1= Almost clear, no thickening; normal to pink coloration; no to minimal focal scaling, scale 2= Mild, just detectable to mild thickening, pink to light red coloration and predominately fine scaling, scale 3= Moderate, clearly distinguishable to moderate thickening; dull to bright red; moderate scaling and scale 4= Severe, severe thickening with hard edges; bright to deep dark red coloration; severe/coarse scaling covering almost all or all lesions. IGA 0/1 response was defined as clear [0] or almost clear [1] with at least a two-category improvement from Baseline.
Time Frame: Week 16
Population: Randomized Set consisted of all randomized study participants. Study participants with an intercurrent event (discontinuation of IMP prior to Week 16) or who had missing data at Week 16 are counted as non-responders (NRI).
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Bimekizumab 320 mg Q4W
Number analyzed (Participants) | 15 | 32
percentage of participants | 0 | 87.5
Statistical Analysis 1: Comparison: Placebo vs Bimekizumab 320 mg Q4W; Test type: Superiority; p < 0.001, Fisher Exact — P-values for the comparison of treatment groups are based on the Fisher's exact test

3. Secondary Outcome: Percentage of Participants With a Psoriasis Area and Severity Index 100 (PASI100) Response at Week 16
Description: The PASI100 response assessments are based on a 100% improvement in the PASI score from Baseline. This is a scoring system that averages the redness, thickness, and scaliness of the psoriatic lesions (on a 0-4 scale), and weights the resulting score by the area of skin involved. Body divided into 4 areas: head, arms, trunk to groin, and legs to top of buttocks. Assignment of an average score for the redness, thickness, and scaling for each of the 4 body areas with a score of 0 (clear) to 4 (very marked). Determining the percentage of skin covered with PSO for each of the body areas and converting to a 0 to 6 scale. Final PASI= average redness, thickness, and scaliness of the psoriatic skin lesions, multiplied by the involved psoriasis area score of the respective section, and weighted by the percentage of the person's affected skin for the respective section. The minimum possible PASI score is 0= no disease, the maximum score is 72= maximal disease.
Time Frame: Week 16
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Bimekizumab 320 mg Q4W
Number analyzed (Participants) | 15 | 32
percentage of participants | 0 | 21.9
Statistical Analysis 1: Comparison: Placebo vs Bimekizumab 320 mg Q4W; Test type: Superiority; p = 0.080, Fisher Exact — P-values for the comparison of treatment groups are based on the Fisher's exact test

4. Secondary Outcome: Percentage of Participants With an Investigator's Global Assessment (IGA) 0 (Clear With at Least 2-category Improvement From Baseline) Response at Week 16
Description: The Investigator's Global Assessment measures the overall psoriasis severity following a 5-point scale (0-4), where scale 0= Clear, no signs of psoriasis; post-inflammatory hyperpigmentation may be present, scale 1= Almost clear, no thickening; normal to pink coloration; no to minimal focal scaling, scale 2= Mild, just detectable to mild thickening, pink to light red coloration and predominately fine scaling, scale 3= Moderate, clearly distinguishable to moderate thickening; dull to bright red; moderate scaling and scale 4= Severe, severe thickening with hard edges; bright to deep dark red coloration; severe/coarse scaling covering almost all or all lesions. IGA 0 response (Clear) is defined as clear [0] with at least a two-category improvement from Baseline.
Time Frame: Week 16
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Bimekizumab 320 mg Q4W
Number analyzed (Participants) | 15 | 32
percentage of participants | 0 | 21.9
Statistical Analysis 1: Comparison: Placebo vs Bimekizumab 320 mg Q4W; Test type: Superiority; p = 0.080, Fisher Exact — P-values for the comparison of treatment groups are based on the Fisher's exact test

5. Secondary Outcome: Percentage of Participants With a Psoriasis Area and Severity Index 75 (PASI75) Response at Week 4
Description: The PASI75 response assessments are based on at least 75% improvement in the PASI score from Baseline. This is a scoring system that averages the redness, thickness, and scaliness of the psoriatic lesions (on a 0-4 scale), and weights the resulting score by the area of skin involved. Body divided into 4 areas: head, arms, trunk to groin, and legs to top of buttocks. Assignment of an average score for the redness, thickness, and scaling for each of the 4 body areas with a score of 0 (clear) to 4 (very marked). Determining the percentage of skin covered with PSO for each of the body areas and converting to a 0 to 6 scale. Final PASI= average redness, thickness, and scaliness of the psoriatic skin lesions, multiplied by the involved psoriasis area score of the respective section, and weighted by the percentage of the person's affected skin for the respective section. The minimum possible PASI score is 0= no disease, the maximum score is 72= maximal disease.
Time Frame: Week 4
Population: Randomized Set consisted of all randomized study participants. Study participants with an intercurrent event (discontinuation of IMP) prior to their Week 4 PASI assessment or who had missing data at Week 4 are counted as non-responders (NRI).
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Bimekizumab 320 mg Q4W
Number analyzed (Participants) | 15 | 32
percentage of participants | 0 | 75.0
Statistical Analysis 1: Comparison: Placebo vs Bimekizumab 320 mg Q4W; Test type: Superiority; p < 0.001, Fisher Exact — P-values for the comparison of treatment groups are based on the Fisher's exact test

6. Secondary Outcome: Percentage of Participants With a Patient Symptom Diary (PSD) (P-SIM) Response for Itch at Week 16
Description: The PSD (P-SIM) was designed for use as a daily diary to collect data about the experience of participants with moderate to severe psoriasis related to the severity of signs, symptoms or impacts, at their worst during the past 24 hours, on a 0-10 point numeric rating scale (NRS) where 0 (no symptoms/impact) and 10 (very severe symptoms/worst impact). It consists of 14 items measuring: redness, scaling, cracking, lesions, thickening, itch, pain, burning, dryness, irritation, sensitivity, fatigue, embarrassment and choice of clothing. A weekly score for each item (including itch) is obtained as an average of daily values for the considered item over the 7 days preceding the visit (weekly score range: 0 (no itch)-10 (very severe itch)). Itch response was defined as a reduction from baseline to Week 16 of at least 4 points on the PSD itch weekly score.
Time Frame: Week 16
Population: Randomized Set consisted of all randomized study participants. The denominator when calculating the percentage of participants with a response to the PSD itch item is the number of participants with a baseline itch score >=4 and the numerator is the number of participants with a PSD response for itch at Week 16. Study participants with an intercurrent event (discontinuation of IMP prior to Week 16) or who had missing data at Week 16 are counted as non-responders (NRI).
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Bimekizumab 320 mg Q4W
Number analyzed (Participants) | 12 | 26
percentage of participants | 0 | 57.7
Statistical Analysis 1: Comparison: Placebo vs Bimekizumab 320 mg Q4W; Test type: Superiority; p < 0.001, Fisher Exact — P-values for the comparison of treatment groups are based on the Fisher's exact test

7. Secondary Outcome: Percentage of Participants With a Patient Symptom Diary (PSD) (P-SIM) Response for Pain at Week 16
Description: The PSD (P-SIM) was designed for use as a daily diary to collect data about the experience of participants with moderate to severe psoriasis related to the severity of signs, symptoms or impacts, at their worst during the past 24 hours, on a 0-10 point NRS where 0 (no symptoms/impact) and 10 (very severe symptoms/worst impact). It consists of 14 items measuring: redness, scaling, cracking, lesions, thickening, itch, pain, burning, dryness, irritation, sensitivity, fatigue, embarrassment and choice of clothing. A weekly score for each item (including pain) is obtained as an average of daily values for the considered item over the 7 days preceding the visit (weekly score range: 0 (no pain)-10 (very severe pain)). Pain response was defined as a reduction from baseline to Week 16 of at least 4 points on the PSD pain weekly score.
Time Frame: Week 16
Population: Randomized Set consisted of all randomized study participants. The denominator when calculating the percentage of participants with a response to the PSD pain item is the number of participants with a baseline pain score >=4 and the numerator is the number of participants with a PSD response for pain at Week 16. Study participants with an intercurrent event (discontinuation of IMP prior to Week 16) or who had missing data at Week 16 are counted as non-responders (NRI).
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Bimekizumab 320 mg Q4W
Number analyzed (Participants) | 10 | 24
percentage of participants | 0 | 62.5
Statistical Analysis 1: Comparison: Placebo vs Bimekizumab 320 mg Q4W; Test type: Superiority; p < 0.001, Fisher Exact — P-values for the comparison of treatment groups are based on the Fisher's exact test

8. Secondary Outcome: Percentage of Participants With a Patient Symptom Diary (PSD) (P-SIM) Response for Scaling at Week 16
Description: The PSD (P-SIM) was designed for use as a daily diary to collect data about the experience of participants with moderate to severe psoriasis related to the severity of signs, symptoms or impacts, at their worst during the past 24 hours, on a 0-10 point numeric rating scale (NRS) where 0 (no symptoms/impact) and 10 (very severe symptoms/worst impact). It consists of 14 items measuring: redness, scaling, cracking, lesions, thickening, itch, pain, burning, dryness, irritation, sensitivity, fatigue, embarrassment and choice of clothing. A weekly score for each item (including scaling) is obtained as an average of daily values for the considered item over the 7 days preceding the visit (weekly score range: 0 (no scaling)-10 (very severe scaling)). Scaling response was defined as a reduction from baseline to Week 16 of at least 4 points on the PSD scaling weekly score.
Time Frame: Week 16
Population: Randomized Set consisted of all randomized study participants. The denominator when calculating the percentage of participants with a response to the PSD scaling item is the number of participants with a baseline scaling score >=4 and the numerator is the number of participants with a PSD response for scaling at Week 16. Study participants with an intercurrent event (discontinuation of IMP prior to Week 16) or who had missing data at Week 16 are counted as non-responders (NRI).
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Bimekizumab 320 mg Q4W
Number analyzed (Participants) | 13 | 28
percentage of participants | 0 | 64.3
Statistical Analysis 1: Comparison: Placebo vs Bimekizumab 320 mg Q4W; Test type: Superiority; p < 0.001, Fisher Exact — P-values for the comparison of treatment groups are based on the Fisher's exact test

9. Secondary Outcome: Percentage of Participants With Scalp IGA Response 0/1 (Clear or Almost Clear With at Least a 2-category Improvement From Baseline) at Week 16 for Study Participants With Scalp Psoriasis (PSO) at Baseline
Description: Participants with scalp involvement at Baseline were defined as those with a scalp IGA score >0 at Baseline. Scalp lesions were assessed in terms of clinical signs of redness, thickness, and scaliness using a 5-point scale (0=Clear, 1=Almost Clear, 2=Mild, 3=Moderate, 4= Severe). Scalp IGA response 0/1 at Week 16 was defined as clear (0) or almost clear (1) with at least a 2-category improvement from Baseline to Week 16.
Time Frame: Week 16
Population: Randomized Set consisted of all randomized study participants. Here, Number of Participants analyzed reflect those with a scalp IGA Baseline score >=2. Study participants with an intercurrent event (discontinuation of IMP prior to Week 16) or who had missing data at Week 16 are counted as non-responders (NRI).
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Bimekizumab 320 mg Q4W
Number analyzed (Participants) | 14 | 29
percentage of participants | 7.1 | 86.2
Statistical Analysis 1: Comparison: Placebo vs Bimekizumab 320 mg Q4W; Odds ratio of scalp IGA response for bimekizumab group compared with placebo group using CMH; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — P-values for the comparison of treatment groups are based on the CMH test from the general association; Odds Ratio (OR) = 81.250, 95% CI 2-sided [8.216 to 803.544]

10. Secondary Outcome: Percentage of Participants With Dermatology Life Quality Index (DLQI) 0/1 Response at Week 16
Description: The DLQI is a skin disease-specific questionnaire aimed at the evaluation of how symptoms and treatment affect study participants' health related quality of life (QOL). This instrument asks study participants about symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment. It has been shown to be valid and reproducible in study participants with PSO. The DLQI total score ranges from 0 to 30, with higher scores indicating lower health related QOL. A 4-point change in the DLQI total score has been reported to be meaningful for the study participant (within-participant minimal important difference); while a DLQI total score of 0 or 1 indicates no impact of the skin disease on participant's life.
Time Frame: Week 16
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Bimekizumab 320 mg Q4W
Number analyzed (Participants) | 15 | 32
percentage of participants | 6.7 | 46.9
Statistical Analysis 1: Comparison: Placebo vs Bimekizumab 320 mg Q4W; Odds ratio of DLQI total score response for bimekizumab group compared with placebo group using CMH; Test type: Superiority; p = 0.007, Cochran-Mantel-Haenszel — P-values for the comparison of treatment groups are based on the CMH test from the general association; Odds Ratio (OR) = 12.353, 95% CI 2-sided [1.447 to 105.443]

11. Secondary Outcome: Percent Change From Baseline in Body Surface Area (BSA) Affected by PSO at Week 16
Description: The Total BSA affected by PSO was entered as a percentage from 0 to 100.
Time Frame: Baseline, Week 16
Population: Randomized Set consisted of all randomized study participants. Study participants with an intercurrent event (discontinuation of IMP prior to Week 16) or who had missing data at Week 16 are imputed using last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Bimekizumab 320 mg Q4W
Number analyzed (Participants) | 15 | 32
percent change | -3.028 (8.926) | -83.472 (6.026)
Statistical Analysis 1: Comparison: Placebo vs Bimekizumab 320 mg Q4W; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -80.444, 95% CI 2-sided [-102.509 to -58.379]

12. Secondary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs) Throughout the Study
Description: An adverse event is any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of IMP, whether or not considered related to the IMP. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of IMP. TEAEs were defined as those AEs that have a start date on or following the first dose of investigational medicinal product (IMP) through the end of the time at risk.
Time Frame: From Baseline to End of Safety Follow-Up (SFU) (up to Week 32)
Population: The Safety Set consisted of all study participants that received at least 1 dose of the IMP.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Bimekizumab 320 mg Q4W
Number analyzed (Participants) | 15 | 32
percentage of participants | 40.0 | 50.0

13. Secondary Outcome: Percentage of Participants With Treatment-emergent Serious Adverse Events (TESAEs) Throughout the Study
Description: A serious adverse event (SAE) is any untoward medical occurrence that at any dose: 1) Results in death 2) Is life-threatening 3) Requires in participant hospitalisation or prolongation of existing hospitalisation 4) Resulted in persistent disability/incapacity 5) Is a congenital anomaly or birth defect 6) Other important medical events which based on medical or scientific judgement may jeopardise the participants, or may require medical or surgical intervention to prevent any of the above.
Time Frame: From Baseline to End of Safety Follow-Up (up to Week 32)
Population: The Safety Set consisted of all study participants that received at least 1 dose of the IMP.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Bimekizumab 320 mg Q4W
Number analyzed (Participants) | 15 | 32
percentage of participants | 6.7 | 0

14. Secondary Outcome: Percentage of Participants With TEAEs Leading to Permanent Discontinuation of Investigational Medicinal Product (IMP) Throughout the Study
Description: An adverse event is any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of IMP, whether or not considered related to the IMP. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of IMP. TEAEs were defined as those AEs that have a start date on or following the first dose of IMP through the end of the time at risk.
Time Frame: From Baseline to End of Safety Follow-Up (up to Week 32)
Population: The Safety Set consisted of all study participants that received at least 1 dose of the IMP.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Bimekizumab 320 mg Q4W
Number analyzed (Participants) | 15 | 32
percentage of participants | 0 | 0

15. Secondary Outcome: Change From Baseline in Patient Health Questionnaire 9 (PHQ-9) at Week 16
Description: The PHQ-9 is a multipurpose instrument for screening, diagnosing, monitoring, and measuring the severity of depression. The PHQ-9 score ranges from 0 to 27 with higher scores indicating a worse state. A score of 5 to 9 is considered to be minimal symptoms of depression. A score of 10 to 14 is considered minor depression, dysthymia, or mild major depression. A score of 15 to 19 is considered to indicate moderately severe major depression, and a score ≥20 is considered to be severe major depression. Change from Baseline is derived as post-Baseline score minus Baseline score, where a positive change indicates worsening and a negative change indicates improvement.
Time Frame: Baseline, Week 16
Population: The Safety Set consisted of all study participants that received at least 1 dose of the IMP. Study participants with missing data at Week 16 were imputed using LOCF.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Bimekizumab 320 mg Q4W
Number analyzed (Participants) | 15 | 32
scores on a scale | -2.1 (5.1) | -2.4 (3.2)

ADVERSE EVENTS:
Time Frame: From Baseline to End of Safety Follow-Up (up to Week 32)
Description: Treatment-emergent AEs (TEAEs) were defined as those AEs that have a start date on or following the first dose of investigational medicinal product (IMP) through the end of the time at risk. TEAEs were analyzed for Safety Set.
Arm/Group | Placebo | Bimekizumab 320 mg Q4W
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/32
Serious Adverse Events (participants affected / at risk) | 1/15 | 0/32
Other Adverse Events (participants affected / at risk) | 6/15 | 11/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=15) | Bimekizumab 320 mg Q4W (N=32)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=15) | Bimekizumab 320 mg Q4W (N=32)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Corona virus infection (Infections and infestations) | 1 (1) | 7 (7)
Tinea pedis (Infections and infestations) | 0 (0) | 2 (2)
Bacteriuria (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Psychiatric evaluation abnormal (Investigations) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
This study protocol was not submitted to FDA, and was not conducted under a US IND or IDE.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-08-16): https://cdn.clinicaltrials.gov/large-docs/49/NCT05020249/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-15): https://cdn.clinicaltrials.gov/large-docs/49/NCT05020249/SAP_001.pdf